CLINICAL TRIAL: NCT05128487
Title: A Phase 1/2, Open-label Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of NDI-101150 Administered as Monotherapy or in Combination With Pembrolizumab in Patients With Solid Tumors
Brief Title: A Study of NDI 1150-101 in Patients With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nimbus Saturn, Inc. (Industry)
Responsible Party: Sponsor
Organization: Nimbus Therapeutics (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1150-101
Record Dates: First submitted 2021-10-22; First posted 2021-11-22 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumor; Renal Cell Carcinoma (Kidney Cancer); Gastric and Gastroesophageal Junction (GEJ) Adenocarcinoma; Non-Small Cell Lung Cancer
Keywords: Dose escalation phase; Dose expansion phase; Hematopoietic progenitor kinase 1; NDI-101150; First-in-human; Maximum tolerated dose; Recommended Phase 2 dose; Renal Cell Carcinoma; Gastric and gastroesophageal junction cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Adenocarcinoma; Carcinoma, Non-Small-Cell Lung; Hereditary Sensory and Autonomic Neuropathies | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NDI-101150 (Monotherapy) (Experimental): Patients in escalation and expansion, will receive NDI-101150 capsules orally once daily continuously in 4-week cycles (28 days).
  Interventions: Drug: NDI-101150
- NDI-101150-Pembrolizumab (Combination therapy) (Experimental): Patients in escalation and expansion phase, will receive NDI-101150 capsules orally once daily continuously in 3-week cycles (21 days), along with pembrolizumab via intravenous (IV) infusion at a dose of 200 mg every 3 weeks.
  Interventions: Drug: NDI-101150; Drug: Pembrolizumab

INTERVENTIONS:
Drug: NDI-101150 — NDI-101150 capsules
Drug: Pembrolizumab — Pembrolizumab IV infusion
  Arms: NDI-101150-Pembrolizumab (Combination therapy)

SUMMARY:
This study is to determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) and to investigate the safety, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of NDI-101150 given as monotherapy or in combination with pembrolizumab in adult patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label, first-in-human, Phase 1/2 study.

The study will consist of 2 phases:

* The Dose Escalation Phase: designed to evaluate the safety and tolerability of NDI-101150 as monotherapy (Arm 1) and in combination with pembrolizumab (Arm 2) in patients with advanced solid tumors.
* The Dose Expansion Phase: designed to evaluate the safety and efficacy of NDI-101150 as monotherapy (Arm 1) and in combination with pembrolizumab (Arm 2) in disease-specific dose expansion cohorts: gastric and gastroesophageal junction [GEJ] cancer, non-small cell lung cancer [NSCLC], and renal cell carcinoma [RCC].

Each phase of the study will consist of 3 periods:

* A Screening period of up to 28 days during which patient eligibility will be reviewed and approved by the Sponsor.
* Treatment period that will extend from Cycle 1 Day 1 until progression of disease (PD), unacceptable toxicity, withdrawal of consent, start of a new systemic anticancer treatment, discontinuation of the patient by the Investigator, or termination of the study by the Sponsor. This will also include Safety Follow-up Visit 30 days [+3 days] after the last dose of investigational medicinal product.
* Post treatment Follow-up period which will continue until lost to follow-up, withdrawal of consent, or the End of the Study (whichever comes first).

ELIGIBILITY:
Key Inclusion Criteria:

* Life expectancy of ≥ 12 weeks
* Measurable or non-measurable disease for Dose Escalation; measurable disease using RECIST v1.1 is required for Dose Expansion
* Recovered from prior therapy to Grade ≤ 1 or return to baseline status (except for alopecia)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients with adequate bone marrow, kidney and liver function
* Last dose of previous anticancer therapy ≥ 4 weeks prior to first dose of NDI-101150; includes prior anti-PD-1 or anti-PD-L1 therapy, other anticancer therapy, radiotherapy, or surgical intervention
* For Dose Escalation Phase Only (Dose Escalation, Monotherapy and Combination Therapy): Histologically or cytologically confirmed advanced or metastatic solid tumors for whom no standard therapies are available or refractory to standard therapy
* For Dose Expansion Phase (Dose Expansion, Monotherapy and Combination Therapy): Willing to consent to required tumor biopsy(ies). Histologically or cytologically confirmed advanced or metastatic G/GEJ, NSCLC or RCC for which no standard therapy is available or are refractory to standard therapy

Key Exclusion Criteria:

* Previous solid organ or hematopoietic cell transplant
* Central nervous system (CNS) malignant disease not previously treated, active leptomeningeal disease, uncontrolled symptomatic CNS involvement, or CNS malignant disease requiring steroid or other therapeutic intervention
* Prior anticancer therapy within 2-6 weeks of trial start (depending on nature of therapy).
* Clinically significant cardiovascular disease
* History of severe hypersensitivity reaction to treatment with monoclonal antibody(ies) (for combination therapy cohorts only)
* History of interstitial lung disease, idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of history of pneumonitis on chest computed tomography scan in the last 6 months
* Known additional malignancy that is active and/or in progression requiring treatment
* Unstable or severe uncontrolled medical condition (e.g., unstable cardiac function, unstable pulmonary condition, uncontrolled diabetes, thromboembolic event within the past 3 months) or any important medical or psychiatric illness or abnormal laboratory finding
* Unable to discontinue medications that are strong inducers or inhibitors of CYP3A4 and/or CYP2C8
* History of severe irAE that led to permanent discontinuation of prior immunotherapy
* History of recent Grade >/= 3 irAE or any Grade 4 life-threatening irAE, neurologic or ocular AE of any grade while receiving prior immunotherapy

NOTE: Other protocol defined Inclusion and Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Part 1: Frequency of dose-limiting toxicities (DLTs) | Cycle 1 (28 days)
Part 2: Objective response rate (ORR) | Up to approximately 34 months

SECONDARY OUTCOMES:
Part 1 and Part 2: Number of patients with adverse events (AEs) and Serious adverse events (SAEs) | From Screening (Day -28 to Day -1) until safety follow-up (>30 days after last dose) [Assessed up to 37 months]
Part 1 and Part 2: Maximum plasma concentration (Cmax) of NDI-101150 | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 1 Day 2, Cycle 2 Day 2 (Monotherapy); at EOT (end-of-treatment)/ET (early termination) [Cycle length is 28 days for monotherapy and 21 days for combination therapy] (Up to 37 months)
Part 1 and Part 2: Time to maximum plasma concentration (tmax) of NDI-101150 | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 1 Day 2, Cycle 2 Day 2 (Monotherapy); at EOT (end-of-treatment)/ET (early termination) [Cycle length is 28 days for monotherapy and 21 days for combination therapy] (Up to 37 months)
Part 1 and Part 2: Area under the concentration-time curve from time zero to the last observable concentration (AUC0-t) of NDI-101150 | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 1 Day 2, Cycle 2 Day 2 (Monotherapy); at EOT (end-of-treatment)/ET (early termination) [Cycle length is 28 days for monotherapy and 21 days for combination therapy] (Up to 37 months)
Part 1 and Part 2: Area under the concentration-time curve extrapolated to infinity (AUC0-∞) of NDI-101150 | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 1 Day 2, Cycle 2 Day 2 (Monotherapy); at EOT (end-of-treatment)/ET (early termination) [Cycle length is 28 days for monotherapy and 21 days for combination therapy] (Up to 37 months)
Part 1: Objective response rate (ORR) | Assessed up to 37 months
Part 1 and Part 2: Progression-free survival (PFS) | From first dose until confirmed progression of disease (PD) or death (Assessed up to 37 months)
Part 1 and Part 2: Duration of response (DOR) | Time from first response until confirmed PD (Assessed up to 37 months)
Part 1 and Part 2: Time to response (TTR) | Time from first dose until first response (Assessed up to 37 months)
Part 2: Overall survival | Assessed up to 37 months

CONTACTS AND LOCATIONS:
Overall Officials: Anita Scheuber, MD, Study Director — Nimbus Saturn
Locations (19):
- United States (19):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Ocala Oncology Center, Ocala, Florida
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Henry Ford Cancer, Detroit, Michigan
  - HealthPartners Cancer Research Center, Saint Paul, Minnesota
  - Washington University, St Louis, Missouri
  - Hackensack University, Hackensack, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Center for Oncology and Blood Disorders, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Oncology, Fairfax, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No